CLINICAL TRIAL: NCT04080583
Title: Short Active Lives Survey in Chronic Lung Conditions: an Exploratory Study
Brief Title: Short Active Lives Survey in Chronic Lung Conditions
Status: Completed | Type: Observational
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Other Study IDs: 190501
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2020-01

CONDITIONS: Lung Diseases
Keywords: Physical activity; Health Status
MeSH Terms: conditions — Lung Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Usual Care: People with a chronic lung condition who are physically inactive

SUMMARY:
Short Actives Lives Survey is a common tool used to measure physical activity in the UK population. Self-reported measures such as the Short Active Lives Survey can be prone to bias. As such, during project evaluations, benefits may be exaggerated due to over-reporting of physical activity or downplayed due to underreporting of physical activity. There is also a lack of research reporting the typical short-term and long-term changes in physical activity (measured by the Short Active Lives Survey) in people with chronic lung conditions who are not receiving support to become active (i.e. usual care, control groups). Accelerometers are small lightweight activity monitors that can be worn on the waist. These monitors are known to provide accurate and reliable objective assessment of physical activity in people with lung conditions.

This research study will recruit a cohort of inactive people with lung conditions and determine changes in physical activity measured by both the Short Active Lives Survey and one of the most valid accelerometers used in people with lung conditions (Actigraph GT3X). The study will also evaluate how these physical activity measures relate to general health (health status and health care use) of people with lung conditions over 12 months. This study will provide information on the usefulness of using the Short Active Lives Survey in the future for measuring physical activity in people with lung conditions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Obstructive Pulmonary Disease, Bronchiectasis, Interstitial Lung Disease, Lung Cancer, Mesothelioma or Asthma
* Physically inactive defined as completing less than 30 minutes ore more of moderate intensity equivalent physical activity per week (measured by the Short Active Lives Survey)

Exclusion Criteria:

* Adults without a diagnosis of Chronic Obstructive Pulmonary Disease, Bronchiectasis, Interstitial Lung Disease, Lung Cancer, Mesothelioma or Asthma
* Age < 18 Years
* Completing 30 minutes or more of moderate intensity equivalent (MIE) physical activity per week
* Inability or unwillingness to sign informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligibility criteria has been designed to be as broad as possible so that findings can be generalisable to the wider population of inactive people with lung conditions. The main study population will be recruited via convenience sampling at the participant identification centres within Lincolnshire Community Health Services, South Lincolnshire CCG, South West Lincolnshire CCG, Lincolnshire East CCG, Lincolnshire West CCG and United Lincolnshire Hospitals NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Minutes of self-reported moderate intensity equivalent physical activity per week | Baseline to 12 months
  Short Active Lives Survey

SECONDARY OUTCOMES:
Accelerometer measured physical activity: time (minutes per day) spent in moderate intensity activity | Baseline to 12 months
  Actigraph wGT3X-BT
Accelerometer measured physical activity: time (minutes per week) spent in light activity | Baseline to 12 months
  Actigraph wGT3X-BT
Accelerometer measured physical activity including: time (minutes per week) spent in vigorous activity | Baseline to 12 months
  Actigraph wGT3X-BT
Accelerometer measured physical activity: time (minutes per day) spent in sedentary state | Baseline to 12 months
  Actigraph wGT3X-BT
Accelerometer measured physical activity: average daily steps | Baseline to 12 months
  Actigraph wGT3X-BT
Accelerometer measured physical activity including: daily vector magnitude units | Baseline to 12 months
  Actigraph wGT3X-BT
EQ5D index | Baseline to 12 months
  Based on self-rating of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension is rated between 1 (no problems) to 5 (unable to/extreme problems). Dimensions are combined to produce a five-digit number describing the individual's health status (ranging from 11111 to 55555). Five digit number converted to an index based on the EQ-5D-5L value set for England. Index ranges from -0.208 (worst possible health) to 1.000 (best possible health).
EQ VAS | Baseline to 12 months
  Self-report of health status on a scale, 0 (worst health) - 100 (best health)
Cost questionnaire | Baseline to 12 months
  NHS resource use questionnaire
Demographics: | Baseline to 12 months
  Age, gender, ethnicity, comorbidities, social deprivation, MRC degree of breathlessness, oxygen use

CONTACTS AND LOCATIONS:
Overall Officials: Arwel W Jones, PhD, Principal Investigator — University of Lincoln
Locations (1):
- University of Lincoln, Lincoln, Lincolnshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No